CLINICAL TRIAL: NCT02239016
Title: Screening Patients With Sickle Cell Disease for Kidney Damage
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Sponsor
Other Study IDs: 2009-0026
Record Dates: First submitted 2014-08-22; First posted 2014-09-12 (Estimated); Last update posted 2021-03-29 (Actual); Status verified 2021-03

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Hgb SS; Hgb SC; Sβ-Thalassemia
MeSH Terms: conditions — Anemia, Sickle Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Urine, whole blood and serum
Oversight: Data Monitoring Committee: No

SUMMARY:
This study aims to study the temporal course of sickle nephropathy and assess novel biomarkers that can predict patients prone to nephropathy.

DETAILED DESCRIPTION:
Sickle cell disease causes kidney damage that gets worse with increasing age, leading to chronic kidney disease and kidney failure in nearly one third of patients with sickle cell disease. Some patients develop kidney damage at a young age and others show mild kidney damage at older ages. We do not know the natural progression of kidney damage in sickle cell disease patients, nor do we know who is more prone to develop severe kidney damage. Therefore, currently, there are no preventative measures or treatments for sickle cell related kidney disease. The purpose of this research study is to collect data that will help in assessing the progression of kidney damage in sickle cell disease, develop novel urine and blood tests that can predict kidney damage early, and developing treatment ideas for intervention and prevention of kidney damage that eventually leads to kidney failure.

ELIGIBILITY:
Inclusion Criteria:

* Sickle cell disease (i.e. Hgb SS, Hgb SC, Sβ-Thalassemia)
* Individuals at baseline/steady state (absence of fever or acute sickle event, defined as vaso-occlusive pain crises, acute chest syndrome, splenic sequestration, stroke, priapism) for three weeks.
* Adult Subjects > 18 years of age: ability to consent to donate blood and/or urine for research purposes only.
* Newborn to < 18 years of age: ability of parent/legal guardian to consent for peripheral blood and/or urine samples to be obtained for research purposes only.

Exclusion Criteria:

* Hematologic malignancy
* Patients that either do not have the ability to undergo the informed consent process or whose parent/legal guardian does not have the ability to undergo the informed consent process

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Sickle cell clinics at various universities and hospitals.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2009-04; Primary Completion 2019-07-29 (Actual); Study Completion 2020-07-29 (Actual)

PRIMARY OUTCOMES:
Rate of progression of microalbuminuria. | Baseline through 36 months

SECONDARY OUTCOMES:
Evaluation of novel urinary biomarkers. | baseline, year 1, year 2 and year 3

CONTACTS AND LOCATIONS:
Overall Officials: Punam Malik, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (4):
- United States (4):
  - Emory University (Children's Healthcare of Atlanta Pediatric Hospital), Atlanta, Georgia
  - Univeristy of Louisville (Kosair Children's Hospital), Louisville, Kentucky
  - National Institutes of Health Clinical Center, Bethesda, Maryland
  - Akron Childen's Hospital, Akron, Ohio

REFERENCES:
- [Result] Sundaram N, Bennett M, Wilhelm J, Kim MO, Atweh G, Devarajan P, Malik P. Biomarkers for early detection of sickle nephropathy. Am J Hematol. 2011 Jul;86(7):559-66. doi: 10.1002/ajh.22045. Epub 2011 May 31. PMID 21630304
- [Derived] Niss O, Lane A, Asnani MR, Yee ME, Raj A, Creary S, Fitzhugh C, Bodas P, Saraf SL, Sarnaik S, Devarajan P, Malik P. Progression of albuminuria in patients with sickle cell anemia: a multicenter, longitudinal study. Blood Adv. 2020 Apr 14;4(7):1501-1511. doi: 10.1182/bloodadvances.2019001378. PMID 32289161